CLINICAL TRIAL: NCT02849496
Title: A Phase II Open-Label, Randomized Study of PARP Inhibition (Olaparib) Either Alone or in Combination With Anti-PD-L1 Therapy (Atezolizumab; MPDL3280A) in Homologous DNA Repair (HDR) Deficient, Locally Advanced or Metastatic Non-HER2-Positive Breast Cancer
Brief Title: Testing Olaparib Either Alone or in Combination With Atezolizumab in BRCA Mutant Non-HER2-positive Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-01130; NCI-2016-01130 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1608018258; 10020 (Other: Yale University Cancer Center LAO); 10020 (Other: CTEP); UM1CA186644 (NIH); UM1CA186686 (NIH); UM1CA186688 (NIH); UM1CA186689 (NIH); UM1CA186691 (NIH); UM1CA186709 (NIH)
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Locally Advanced Unresectable Breast Carcinoma; Metastatic Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — atezolizumab; Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; olaparib; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (olaparib) (Experimental): Patients receive olaparib PO BID on days 1-21 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression may cross-over to Arm II. Patients undergo an x-ray, CT scan, MRI, bone scan, and/or PET scan as well as a biopsy and blood sample collection throughout the trial. Patients may also undergo a bone marrow aspiration and biopsy on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Olaparib; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Procedure: X-Ray Imaging
- Arm II (olaparib, atezolizumab) (Experimental): Patients receive olaparib as in Arm I and atezolizumab IV over 30-60 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo an x-ray, CT scan, MRI, bone scan, and/or PET scan as well as a biopsy and blood sample collection throughout the trial. Patients may also undergo a bone marrow aspiration and biopsy on study.
  Interventions: Drug: Atezolizumab; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Olaparib; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Procedure: X-Ray Imaging

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
  Arms: Arm II (olaparib, atezolizumab)
Procedure: Biopsy Procedure — Undergo a biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Bone Scan — Undergo a bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo a CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281
Procedure: Positron Emission Tomography — Undergo a PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Questionnaire Administration — Ancillary studies
Procedure: X-Ray Imaging — Undergo an x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This randomized phase II trial studies how well olaparib with or without atezolizumab work in treating patients with non-HER2-positive breast cancer that has spread to nearby tissue or lymph nodes (locally advanced), that cannot be removed by surgery (unresectable), or that has spread from where it first started (primary site) to other places in the body (metastatic). Olaparib is an inhibitor of PARP, an enzyme that helps repair deoxyribonucleic acid (DNA) when it becomes damaged. Blocking PARP may help keep cancer cells from repairing their damaged DNA, causing them to die. PARP inhibitors are a type of targeted therapy. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the tumor, and may interfere with the ability of tumor cells to grow and spread. It is not known whether giving olaparib with or without atezolizumab will work better in patients with non-HER2-positive breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the progression free survival (PFS) between two study arms, i.e., olaparib monotherapy (arm 1) and olaparib + atezolizumab in combination (arm 2) based on normal Response Evaluation Criteria in Solid Tumors (RECIST) criteria in patients with locally advanced or metastatic non-HER2-positive breast cancer harboring homologous deoxyribonucleic acid (DNA) repair (HDR) through BRCA 1/2 mutation.

SECONDARY OBJECTIVES:

I. To compare the progression free survival (PFS) between the two study arms based on immune response criteria.

II. To compare the time to treatment failure (TTF) between the two study arms based on immune response criteria and normal RECIST.

III. To compare the overall response rate (ORR) between the two study arms based on immune response criteria and normal RECIST.

IV. To compare the duration of response (DoR) between the two study arms based on immune response criteria and normal RECIST.

V. Determine the changes in extent of mutational burden in BRCA 1/2 mutated tumors at baseline and at progression.

VI. Evaluate and characterize changes in the extent of PD-L1 expression and tumor immune infiltrates.

VII. Retrospectively evaluate tumors with limited immune infiltrate (e.g. "non-inflamed") to determine if PARPi increased immune infiltration.

VIII. Determine the immune-related best overall response (irBOR) of olaparib in combination with atezolizumab in locally advanced or metastatic non-HER2+ breast cancer harboring HDR through BRCA 1/2 mutation.

EXPLORATORY OBJECTIVES:

I. Evaluate changes in candidate neoantigen profiles and immune/inflammation signatures using DNA and ribonucleic acid (RNA)-sequencing in serial tumor biopsies.

II. Evaluate and characterize circulating tumor DNA (ctDNA) and immune parameters in blood.

III. Test the hypothesis that DNA repair status affects the tumor-immune interaction.

IV. Characterize mechanism of action of the PARP inhibitor olaparib. V. To explore the inclusion of patient reported symptomatic adverse events. VI. To use anti-Kynurenine antibodies for immunohistochemistry (IHC) as well as unbiased metabolome studies on plasma to understand the metabolic consequences of PARP-inhibition and their effects on immune infiltrates.

VII. To explore pharmacodynamic transcriptional changes induced by treatment in different immune cell populations and with high resolution in single cell RNA sequencing of peripheral blood mononuclear cell (PBMC) preparations. This will also be used to study changes in specific T-cell clonotypes.

VIII. To examine increased mitotic errors during response that are surveilled by the innate immune system.

IX. To test whether mutations or expression changes in genes tied to DNA repair regulation arise during acquired resistance and can be discerned by comparative genomics of pre- and at- progression biopsies.

X. To examine whether biomarker development tied to mitotic errors will be of future utility in predicting PARPi response.

XI. To test DNA methylation relationship to resistance mechanism and RNA sequencing (seq).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive olaparib orally (PO) twice daily (BID) on days 1-21 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression may cross-over to Arm II. Patients undergo an x-ray, computed tomography (CT) scan, magnetic resonance imaging (MRI), bone scan, and/or positron emission tomography (PET) scan as well as a biopsy and blood sample collection throughout the trial. Patients may also undergo a bone marrow aspiration and biopsy on study.

ARM II: Patients receive olaparib as in Arm I and atezolizumab intravenously (IV) over 30-60 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo an x-ray, CT scan, MRI, bone scan, and/or PET scan as well as a biopsy and blood sample collection throughout the trial. Patients may also undergo a bone marrow aspiration and biopsy on study.

After completion of study treatment, patients are followed up at 30 days. Patients who come off treatment for reasons other than disease progression are followed every 4-8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically documented unresectable locally advanced or metastatic non-HER2-positive breast cancer and a known BRCA 1/2 mutation present; both germline and somatic mutations are acceptable, however somatic mutations must be identified by either tumor sequencing of tumor tissue or ctDNA in plasma; patients with BRCA mutations of unknown significance are not allowed
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) by chest x-ray or as >= 10 mm (>= 1 cm) with CT scan, MRI, or calipers by clinical exam
* Prior chemotherapy is allowed, including platinum therapy; patients must not have received chemotherapy for 4 weeks prior to the initiation of study treatment and must have recovery =< grade 1 from any adverse events from any prior chemotherapy (other than alopecia); patients must not have had nitrosoureas or mitomycin C for 6 weeks prior to the initiation of study treatment
* Prior radiation therapy is allowed; patients must not have received minimal radiation therapy (=< 5% of their total marrow volume) within 3 weeks prior to the initiation of study treatment; otherwise, patients must not have received radiation therapy (> 5% of their total marrow volume) within 4 weeks prior to the initiation of study treatment; patients who have received prior radiation to 50% or more of their total marrow volume will be excluded
* Patients who have received prior treatment with anti-CTLA-4 may be enrolled, provided the following requirements are met: minimum of 12 weeks from the first dose of anti-CTLA-4 and > 6 weeks from the last dose, and no history of severe immune-related adverse effects from anti-CTLA-4 (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] grade 3 and 4)
* Treatment with systemic immunosuppressive medications (including, but not limited to, prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) is allowed, provided the following is met: minimum of 2 weeks prior to cycle 1, day 1; patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled; the use of corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
* Prior treatment with systemic immunostimulatory agents (including, but not limited to, interferon [IFN]-alpha or interleukin [IL]-2) is allowed, provided the following is met: minimum of 4 weeks or 5 half-lives of the drug (whichever is longer) prior to cycle 1, day 1
* Patients taking bisphosphonate therapy for symptomatic hypercalcemia are NOT allowed; use of bisphosphonate therapy for other reasons (e.g., bone metastasis or osteoporosis) is allowed
* Prior hormone therapy is allowed; patients must not have received hormone therapy for breast cancer for 2 weeks prior to the initiation of study treatment and must have recovery =< grade 1 from any adverse events related to these therapies (other than alopecia)
* Prior experimental (non-Food and Drug Administration [FDA] approved) therapies and immunotherapies are allowed; patients must not have received these therapies for 4 weeks prior to the initiation of study treatment and must have recovery =< grade 1 from any adverse events of these therapies (other than alopecia); prior treatment with any PARP inhibitor or any anti-PD-1/anti-PD-L1 antibody is NOT allowed
* Other therapies (e.g. targeted therapy such as cyclin-dependent kinase [CDK] inhibitors): patients should have recovered to =< grade 1 drug related toxicity; they must have completed therapy for either a total of duration equivalent to 5 half-lives of the drug or 28 days, whichever is shorter
* Age >= 18 years. No dosing or adverse event data are currently available on the use of olaparib in combination with atezolizumab in patients < 18 years of age; hence, children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 6 months
* Absolute neutrophil count >= 1,500/mcL
* Leukocytes >= 3,000/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 8 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (however, patients with known Gilbert disease who have serum bilirubin level =< 3 x ULN may be enrolled)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x upper limit of normal (ULN) if no liver metastasis; =< 5 x upper ULN if liver metastasis present
* Alkaline phosphatase =< 2.5 x ULN (=< 5 x ULN for patients with documented liver involvement or bone metastases)
* Creatinine clearance >= 51 mL/min/1.73 m^2 by Cockcroft-Gault
* International normalized ratio (INR) and activated partial thromboplastin time (aPTT) =< 1.5 x ULN (this applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation, such as low-molecular-weight heparin or warfarin, should be on a stable dose)
* No features suggestive of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) on peripheral blood smear when performed as clinically indicated
* Patients must have tumors determined to be easily accessible for biopsy and must be willing to have serial biopsies (with a third biopsy upon evidence of disease progression)
* Administration of atezolizumab and/or olaparib may have an adverse effect on pregnancy and poses a risk to the human fetus, including embryo-lethality; women of child-bearing potential and men must agree to use highly effective contraception prior to study entry, for the duration of study participation, and for at least 5 months (150 days) after the last dose of study agent; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use two highly effective forms of contraception in combination prior to the study, for the duration of study participation, and for at least 5 months (150 days) after completion of atezolizumab and/or olaparib administration; women of child-bearing potential: negative serum pregnancy test within 14 days of study treatment and confirmed prior to treatment on day 1; postmenopausal or evidence of non-childbearing status for women of childbearing potential; postmenopausal is defined as:

  * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
  * Luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the post-menopausal range for women under 50
  * Radiation-induced oophorectomy with last menses > 1 year ago
  * Chemotherapy-induced menopause with > 1 year interval since last menses
  * Surgical sterilization (bilateral oophorectomy or hysterectomy)
* Ability to understand and the willingness to sign a written informed consent document
* Subject is able to swallow and retain oral medication and does not have uncontrolled emesis or gastrointestinal disorders likely to interfere with absorption of the study medication
* Patients crossing over from monotherapy to combination therapy do not have to be fully rescreened, as they would have just had tumor assessments and would already have had baseline electrocardiographies (ECGs), etc; however, they do need to meet performance status, organ function, and blood parameters and not meet any of the exclusion criteria
* Patients positive for human immunodeficiency virus (HIV) are NOT excluded from this study, but HIV-positive patients must have:

  * A stable regimen of highly active anti-retroviral therapy (HAART)
  * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
  * A CD4 count above 250 cells/mcL and an undetectable HIV viral load on standard polymerase chain reaction (PCR)-based test

Exclusion Criteria:

* Patients with prior allogeneic bone marrow transplantation, double umbilical cord blood transplantation (dUCBT) or prior solid organ transplantation
* Patients with known brain metastases should be excluded from this clinical trial except as those described below, because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Patients with known primary central nervous system (CNS) malignancy or symptomatic CNS metastases are excluded, with the following exceptions:

  * Patients with asymptomatic untreated CNS disease may be enrolled, provided all of the following criteria are met:

    * Evaluable or measurable disease outside the CNS
    * No metastases to brain stem, midbrain, pons, medulla, cerebellum, or within 10 mm of the optic apparatus (optic nerves and chiasm)
    * No history of intracranial hemorrhage unless it is confined within a lesion previously noted and secondary to gamma knife or another equivalent radiologic therapeutic
    * No history of spinal cord hemorrhage
    * No ongoing requirement for dexamethasone for CNS disease; patients on a stable dose of anticonvulsants are permitted
    * No neurosurgical resection or brain biopsy within 28 days prior to cycle 1, day 1
  * Patients with asymptomatic treated CNS metastases may be enrolled, provided all the criteria listed above are met as well as the following:

    * Radiographic demonstration of improvement upon the completion of CNS directed therapy and no evidence of interim progression between the completion of CNS directed therapy and the screening radiographic study
    * No stereotactic radiation or whole-brain radiation within 28 days prior to cycle 1, day 1
    * Screening CNS radiographic study >= 4 weeks from completion of radiotherapy and >= 2 weeks from discontinuation of corticosteroids
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to olaparib and atezolizumab; patients with a known hypersensitivity to olaparib or any of the excipients of the product
* Prior treatment with any PARP inhibitor or any anti-PD-1/anti-PD-L1 antibody
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease

  * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA
* History or risk of autoimmune disease, including, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, lichen sclerosis, or glomerulonephritis

  * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible
  * Patients with controlled type 1 diabetes mellitus on a stable insulin regimen may be eligible
  * Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

    * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
    * Rash must cover less than 10% of body surface area (BSA)
    * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alclometasone dipropionate 0.05%)
    * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan; history of radiation pneumonitis in the radiation field (fibrosis) is permitted if recovered
* Major surgical procedure within 28 days prior to cycle 1, day 1 and patients must have recovered from any effects of any major surgery; anticipation of need for a major surgical procedure during the course of the study
* Administration of a live, attenuated vaccine within 4 weeks before cycle 1, day 1 or anticipation that such a live, attenuated vaccine will be required during the study and up to 5 months after the last dose of atezolizumab

  * Influenza vaccination should be given during influenza season only (approximately October to March); patients must not receive live, attenuated influenza vaccine within 4 weeks prior to cycle 1, day 1 or at any time during the study
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection; examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, unstable spinal cord compression, superior vena cava syndrome, symptomatic congestive heart failure, unstable angina pectoris, extensive interstitial bilateral lung disease on high resolution computed tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent and would limit compliance with study requirements
* Pregnant women are excluded from this study because olaparib and atezolizumab have the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with olaparib and atezolizumab, breastfeeding should be discontinued if the mother is treated with olaparib and atezolizumab
* Any prior grade >= 3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE > grade 1
* Patients with active seizures or a history of uncontrolled seizure disorder, including focal or generalized seizure within the past year
* Patients requiring treatment with a RANKL inhibitor (e.g. denosumab) who cannot discontinue it before treatment with atezolizumab
* Resting ECG with corrected QT (QTc) > 470 msec or family history of long QT syndrome
* Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil); the required washout period prior to starting olaparib is 2 weeks; because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated drug information reference; medical reference texts such as the Physicians' Desk Reference may also provide this information; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Concomitant use of known strong (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's wort) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil); the required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents; because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated drug information reference; medical reference texts such as the Physicians' Desk Reference may also provide this information; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2017-03-30 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Time measured from randomization, assessed up to 7 years
  The study arms will be compared for duration of response survival with Kaplan-Meier estimates and log-rank tests. The Rothman confidence interval (CI), which is based on Greenwood's variance, Thomas and Grunkemeier CI, and the simultaneous confidence bands by Nair and Hall and Wellner, will be reported. In addition, the possible risk factors will be compared for survival with log-rank test. For multivariate analysis, the proportional hazards Cox model will be applied to investigate potential prognostic factors, such as age and stage of disease of the PFS data. The adjusted p-values of the hazard ratios and the adjusted 95% confidence interval will be reported.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 7 years
  Evaluated by immune response criteria and normal Response Evaluation Criteria in Solid Tumors criteria. The ORR will be estimated using the 95% CI based on Wilson's method. The Fisher's exact test will be applied to examine the difference between two arms. The Wilcoxon rank sum test and Fisher's exact test will be applied to study the association between the response status and the continuous and categorical variables, respectively. The generalized non-linear model and logistic regression will be applied for multivariable data analysis. The adjusted p-value and 95% CI of the odds ratios (OR) will be reported.
Duration of response (DoR) | Time from documentation of tumor response to disease progression, assessed up to 7 years
  The study arms will be compared for duration of response survival with Kaplan-Meier estimates and log-rank tests. The Rothman CI, which is based on Greenwood's variance, Thomas and Grunkemeier CI, and the simultaneous confidence bands by Nair and Hall and Wellner, will be reported. In addition, the possible risk factors will be compared for survival with log-rank test. For multivariate analysis, the proportional hazards Cox model will be applied to investigate potential prognostic factors, such as age and stage of disease of the DoR data. The adjusted p-values of the hazard ratios and the adjusted 95% confidence interval will be reported.

OTHER OUTCOMES:
Change in level of tumor infiltrating lymphocytes (TILs) | Baseline up to 7 years
  Differences between groups will be statistically tested using t-test or Wilcoxon rank sum test for continuous variables (quantitative multiplexed TIL scores) and chi-square test or Fisher's exact test for categorical variables (positive/negative using hematoxylin & eosin). Linear and non-linear restricted cubic spline regression coefficients will also be calculated to determine the association between TIL subtypes in the quadriplegia index of function (QIF) evaluation using continuous scores.
Changes of biomarkers expression using deoxyribonucleic acid (DNA) and ribonucleic acid (RNA)-sequencing | Baseline to up to 7 years
  Will be analyzed using Lasso-based elastic net method. The elastic net method is a variable selection procedure by L1 and L2 penalized estimation that enforces variable selection and shrinkage simultaneously. The penalty parameter that controls the shrinkage of fixed terms and the variable selection will be determined by k-fold cross validation. The statistical analyses will be completed by either R 3.2.1 or statistical analysis system (SAS) 9.4 statistical program in this project.
Changes in extent of mutational burden in BRCA1/2 | Baseline to up to 7 years
  Will be analyzed using Lasso-based elastic net method. The elastic net method is a variable selection procedure by L1 and L2 penalized estimation that enforces variable selection and shrinkage simultaneously. The penalty parameter that controls the shrinkage of fixed terms and the variable selection will be determined by k-fold cross validation. The statistical analyses will be completed by either R 3.2.1 or SAS 9.4 statistical program in this project.
Change in PD-L1 | Baseline to up to 7 years
  Will be analyzed using Lasso-based elastic net method. The elastic net method is a variable selection procedure by L1 and L2 penalized estimation that enforces variable selection and shrinkage simultaneously. The penalty parameter that controls the shrinkage of fixed terms and the variable selection will be determined by k-fold cross validation. The statistical analyses will be completed by either R 3.2.1 or SAS 9.4 statistical program in this project.
Change in PARPi | Baseline to up to 7 years
  Will be analyzed using Lasso-based elastic net method. The elastic net method is a variable selection procedure by L1 and L2 penalized estimation that enforces variable selection and shrinkage simultaneously. The penalty parameter that controls the shrinkage of fixed terms and the variable selection will be determined by k-fold cross validation. The statistical analyses will be completed by either R 3.2.1 or SAS 9.4 statistical program in this project.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M LoRusso, Principal Investigator — Yale University Cancer Center LAO
Locations (58):
- United States (58):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Farmington Health Center, Farmington, Utah
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah

REFERENCES:
- See also: Related Info — https://grants.nih.gov/policy/sharing.htm